CLINICAL TRIAL: NCT01770808
Title: A Randomised, Double-blind, Placebo-controlled Study to Determine if Aquamin (as AquaCal and AquaPT) Improves Digestive Discomfort in Healthy Subjects
Brief Title: A Study to Determine if Aquamin (as AquaCal and AquaPT) Improves Digestive Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Marigot Ltd. (Industry)
Responsible Party: Principal Investigator, Andrea Doolan, Human Studies Manager, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC027
Record Dates: First submitted 2012-05-14; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Digestive System Disorders
Keywords: Bloating; Flatulence; Stomach discomfort
MeSH Terms: conditions — Digestive System Diseases; Flatulence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AquaCal (Experimental): AquaCal is produced by Marigot Ltd. The daily dose of 4 capsules of AquaCal provide 800mg calcium, (the EU RDA for calcium) and 74 mgs Magnesium (EU RDA 375mg).
  Interventions: Dietary Supplement: AquaCal
- AquaPT (Experimental): AquaPT are produced by Marigot Ltd. The daily dose of 4 capsules of AquaPT provides 720mg calcium, 200mgs green tea (polyphenols) and 50 mgs pine bark extract.
  Interventions: Dietary Supplement: AquaPT
- Placebo (Placebo Comparator): Produced by Marigot Ltd
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AquaCal — AquaCal is produced by Marigot Ltd. The daily dose of 4 capsules of AquaCal provide 800mg calcium, (the EU RDA for calcium) and 74 mgs Magnesium (EU RDA 375mg). Subjects swallowed 4 capsules/day for six weeks.
  Arms: AquaCal
Dietary Supplement: AquaPT — AquaPT is produced by Marigot Ltd according to EU and FDA requirements. The daily dose of 4 capsules of AquaPT provides 720mg calcium, 200mgs green tea (polyphenols) and 50 mgs pine bark extract. Subjects swallowed 4 capsules/day for six weeks.
  Arms: AquaPT
Dietary Supplement: Placebo — Subjects swallowed 4 capsules/day for six weeks.
  Arms: Placebo

SUMMARY:
Digestive discomfort includes gastrointestinal symptoms such as abdominal pain, altered bowel habit, flatulence and bloating and can sometimes result from slower intestinal transit and other digestive irregularities.

The objective of this study is to investigate the effect of consuming Aquamin (as AquaCal and AquaPT) on digestive discomfort and symptoms amongst adults without diagnosed gastrointestinal disorders.

DETAILED DESCRIPTION:
Digestive discomfort includes gastrointestinal symptoms such as abdominal pain, altered bowel habit, flatulence and bloating and can sometimes result from slower intestinal transit and other digestive irregularities. Digestive discomfort may lead to health issues in the long-term. In a recent survey of over 1,000 women in the UK, 88% reported having experienced digestive discomfort from time to time, but the majority of them (70%) had never consulted a doctor or nurse. Digestive discomfort is often a source of embarrassment for people; they therefore may be reluctant to address these issues with a healthcare professional.

Aquamin is a seaweed-derived mineral source, which is rich in calcium, magnesium and 74 other trace minerals including zinc, iron and selenium. It is produced from the red algae, Lithothamnion Calcareum, which is found in just three locations in the world, including the south-west coast of Ireland and Iceland. During a five-year life span, these algae absorb essential minerals from the sea - this gives Aquamin its unique multimineral content. The algae then break down naturally and settle on the sea bed. These calcified skeletal remains are harvested, washed, dried and milled and provided in a capsule formulation. Aquamin is proven to deliver digestive health benefits. In a recent study, mice feed on a high-fat 'Western-style' diet (HFWD) and Aquamin, suppressed colon polyp formation and a reduction in systemic inflammatory changes in comparison to those not receiving Aquamin.

The objective of this study is to investigate the effect of consuming Aquamin (as AquaCal and AquaPT) on digestive discomfort and symptoms amongst adults without diagnosed gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be able to give written informed consent.
2. Be a female between 18 and 65 years of age.
3. Be a non-pregnant female.
4. Be in generally good health as determined by the investigator.
5. Have no evidence of gastrointestinal disease or of a functional gastrointestinal disorder as determined by the Bowel Disease Questionnaire.
6. Experience occasional bloating and stomach discomfort, defined as 1-2 times/weeks, but not greater that 2 times/week over the last 3 months.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 18 and greater than 65 years of age.
2. Are pregnant females.
3. Are currently taking probiotics, vitamin supplements or plant sterols ester supplements or have taken them in the past 14 days.
4. Have received a diagnosis or attending a doctor for Irritable Bowel Syndrome or a functional bowel disorder.
5. Experience bloating, flatulence and stomach discomfort greater that 2 times/week, over the last 3 months.
6. Have a significant acute or chronic coexisting illness (cardiovascular, gastrointestinal, endocrinological, immunological, metabolic or any condition which contraindicates, in the investigators judgement, entry to the study).
7. Prior gastrointestinal surgery (apart from appendicectomy and hernia repair) or recent unexplained bleeding.
8. Having a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include anti-inflammatory drugs, corticosteroids, laxatives, enemas, antibiotics (within 1 month), probiotics, anti-coagulants, vitamin supplements and over-the counter non-steroidal analgesics.
9. Be a smoker
10. Suffer from alcohol abuse.
11. Suffer from psychiatric disease.
12. Subjects are lactose intolerant or have dietary habits (slimming or vegetarian diet) which could interfere with the assessment of the study product.
13. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
14. Subjects may not be receiving treatment involving experimental drugs.
15. If the subject has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
16. Have a malignant disease or any concomitant end-stage organ disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change digestive discomfort symptoms at 6 weeks | wk 0 & wk 6
  Global symptom questionnaire

SECONDARY OUTCOMES:
Change abdominal bloating at 6 weeks | Week 0 & 6
  Global symptom questionnaire
Change in flatulence at 6 weeks | Weeks 0 & 6
  Global symptom questionnaire
Change in tummy discomfort at 6 weeks | Weeks 0 & 6
  Global symptom questionnaire
Change in at Cytokines 6 weeks | Weeks 0 & 6
  Plasma cytokines IL6 & IL8

CONTACTS AND LOCATIONS:
Overall Officials: Eamonn Quigley, MD, Principal Investigator — University College Cork
Locations (1):
- Cork University Hospital, Cork, Ireland